CLINICAL TRIAL: NCT03280511
Title: Adjuvant Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) in Resected High Risk Colon Cancer Patients - The PIPAC-OPC3 CC Trial
Brief Title: Adjuvant Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) in Resected High Risk Colon Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Bau Mortensen (Other)
Responsible Party: Sponsor-Investigator, Michael Bau Mortensen, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PIPAC-OPC3
Record Dates: First submitted 2017-09-03; First posted 2017-09-12 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Peritoneum Cancer; Peritoneal Carcinomatosis; Peritoneal Metastases; Colo-rectal Cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Colonic Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Non-randomized, non-blinded phase 2 cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Eligible candidates will be enrolled according to in-/exclusion criteria. Two months after colon resection or immediately after adjuvant chemotherapy (if indicated), a standard laparoscopy including peritoneal lavage, peritoneal biopsies and PIPAC treatment with oxaliplatin 92 mg/m2 will be planned. This procedure will be repeated after another 5 weeks. Follow up CTs after 12, 24 and 36 months will be planned.
  Interventions: Drug: PIPAC

INTERVENTIONS:
Drug: PIPAC — PIPAC is performed during a standard laparoscopy with a capnoperitoneum of 12 mmHg. During PIPAC, oxaliplatin 46 mg/m2 in 150 ml dextrose will be intraperitoneally nebulized at a rate of 0.5 ml/s with a maximum pressure of 200 PSI. The intraperitoneal air will be evacuated after 30 minutes of simple diffusion
  Other Names: Oxaliplatin

SUMMARY:
In this study, patients will be offered two Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) treatments with oxaliplatin after primary resection and standard adjuvant chemotherapy (if indicated) for colon cancer. Furthermore, the study will explore, whether it is possible to find free intraperitoneal tumor cells (FITC) after resection and adjuvant chemotherapy for colon cancer.

DETAILED DESCRIPTION:
In 2015, 3500 patients were diagnosed with colon cancer in Denmark (DCCG Årsrapport 2015, www.dccg.dk). Despite curative intended surgery and perioperative chemotherapy in colon cancers, relapse is often encountered, and across tumor stage recurrence is found in 18-26% of the resected patients. Eighty-six percent of the recurrences are diagnosed within three years after resection, and 36% of the recurrences are diagnosed within the first year regardless of tumor stage. The route of dissemination varies with different cancer types, but a common denominator is the risk of peritoneal metastases (PM). PM is the second most common site of recurrence in colon cancer patients, and accounts for 25-35% of all recurrences. Patients with PM - both in the synchronous and metachronous setting - will often have a very short life expectancy and traditionally, treatment have been nihilistic due to poor performance status and response rates, and most patients with recurrence to the peritoneum will only be treated with best supportive care. During the last two decades, more aggressive treatment strategies have been implemented, including extensive surgery (Cytoreductive surgery, CRS) followed by hyperthermic intraperitoneal chemotherapy (HIPEC). However, CRS and HIPEC are only used in selected patients with limited PM. High risk factors for relapse with PM have been identified, and patients with T4 colon cancers have a risk of relapse with metachronous PM between 12-50%, while patients with intraperitoneally perforated colorectal cancers relapse with PM in 14- 58% of the cases. The risk of metachronous PM in perforated or T4 colorectal cancers has been validated and this is widely recognized in the ongoing trials around Europe, where adjuvant HIPEC is being investigated in patients with high-risk colon tumors to prevent metachronous PM (www.clinicaltrials.gov NCT02231086, NCT02965248, NCT02614534, NCT02974556, NCT01226394).

In addition to tumor stage, free intraperitoneal tumor cells (FITC) are perceived as a precursor of PM, and it is expected, that patients with perforated/T4 colon cancers will have FITC prior to visible recurrence with PM. However, despite the reported impact on the risk of recurrence and poor survival data, the presence of FITC is not routinely investigated, and this may be due to the lack of treatment options regarding the eradication of free tumor cells. In a systematic review of resected patients with stage I-IV colorectal cancer, 13.7% had FITC detected during perioperative peritoneal lavage. The rate of FITC increased with increasing T-stage and the patients with FITC had a significantly increased risk of both local and overall recurrence, plus a significantly increased mortality risk.

Based on the above-mentioned rate of recurrences after resection of high-risk colon cancers and the limited treatment options, new treatment strategies are needed. A German research group has invented a new intraperitoneal chemotherapy delivery method, where the chemotherapy is nebulized within the pressurized abdominal cavity - Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC).

PIPAC As blood supply to the peritoneal surface is scarce, systemic chemotherapy has limited access to the peritoneal cavity, especially when the primary tumor including its exfoliating surface has been resected. Even though intraperitoneal chemotherapy would seem like a tempting alternative, convincing results are still missing. Temperature and pressure are important factors during absorption of fluid from the peritoneal cavity, and the use of a relative low intraperitoneal pressure (2-6 mmHg) seems to increase the inflow of intraperitoneal fluid into the abdominal wall. Studies have confirmed that higher tissue concentrations of chemotherapy may be obtained by increasing the intraperitoneal pressure. After years of extensive testing, and the development of a CE-certified nebulizer (CapnoPen, Capnomed, Villingendorf, Germany) for safe aerosol infusion, a German research group has designed a system that allows a laparoscopy controlled delivery of Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC). The aerosol technique ensures that the entire peritoneal surface is covered by chemotherapy, and this is relevant when trying to eradicate (all) free intraperitoneal tumor cells. With the nebulizer positioned through a standard trocar pointing away from the bowels, a commercially available injection pump (MEDRAD Salient Dual Contrast Injector, Bayer HealthCare, Leverkusen, Germany) provides the necessary pressure to induce an aerosol mist covering the peritoneal cavity. After five minutes, the chemotherapy has been delivered, and the injector is turned off. After an additional 25 minutes of simple diffusion, the aerosol is gone and the remaining intraabdominal CO2 is evacuated through a standard trocar.

PIPAC is safe, both for patients and healthcare workers, and preliminary data suggest encouraging objective tumor response and survival data. Based on the results of the German research group, PIPAC has been implemented at Odense University Hospital in a feasibility and safety study (www.clinicaltrial.gov NCT02320448, The Regional Scientific Ethical Committees for Southern Denmark Project-ID: S-20140211). Accrual has stopped, as the planned 35 patients have been included. 130 PIPAC treatments have been performed so far, and three patients are still in treatment. Preliminary data suggest a good safety profile, both in terms of patient safety and occupational health safety, as demonstrated on The First Scandinavian PIPAC Symposium, April 20th 2017. In brief, environmental and biological analyses demonstrated no risk of chemotherapy exposure to the health care workers, the planned procedures could be completed in 100% of the patients and 90% were discharged within the first postoperative day (range 1-4). In 20% of the procedures using oxaliplatin, the patients had postoperative urinary retention relieved by a singleuse catheter and in less than 5% of the procedures, a serious adverse event (CTCAE grade 3) was encountered (1 small bowel perforation, 1 small bowel obstruction, 1 cholestasis, 1 diarrhea), and there was no mortality.

Detection of FITC FITC is usually detected by analysing smears of sediment from the peritoneal lavage fluid collected during a staging laparoscopy or during the course of surgery. As FITC is routinely investigated in especially Asian gastric cancer patients, the current experience on the detection of FITC arises from studies in gastric cancer patients. A recent meta-analysis described the risk of peritoneal recurrence of gastric cancer, based on analysis of peritoneal lavage fluid. In this study, peritoneal lavage cytology predicted peritoneal recurrence with a sensitivity of only 0.45, while the specificity was 0.92-0.98. By the detection of carcinoembryonic antigen (CEA) in the peritoneal lavage fluid, the sensitivity was 0.77 and the specificity 0.89, whereas the analysis of CEA mRNA raised the sensitivity to 0.87, with a specificity of 0.80. In a systematic review, peritoneal lavage cytology predicted peritoneal recurrence of gastric cancer patients with a sensitivity of 0.11-0.80 and a specificity of 0.86-1.00. By analysing the lavage fluid with immunoassays, immunohistochemistry or Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) mainly towards CEA, the sensitivity and specificity still varied significantly (sensitivity 0.23-1.00, specificity 0.81-0.98). Despite the variable results, the included studies of this systematic review confirmed a significantly reduced median overall survival in patients with FITC. However, there is no standard definition of the techniques or cut off points used to detect FITC - neither in gastric/GEJ cancer patients nor in colon cancer patients.

Study rationale As PIPAC seems to have an effect on visible PM in colon cancer patients, the investigators hypothesize that PIPAC can minimize the risk of PM recurrence in resected high risk colon cancer patients.

Furthermore, the investigators expect that PIPAC can eradicate FITC in these patients.

Study population Danish patients with colon cancer are eligible candidates according to the inclusion criteria. The patients will be included after resection and, if indicated, adjuvant systemic chemotherapy. While expected accrual is based on the number of resected patients at Odense University Hospital, this study will include patients nationwide.

In 2015, 284 patients were resected due to colon cancer at Odense University Hospital (OUH). Ninety-three percent of the resections were with curative intent (n=264), and eighteen percent had T4 tumors (DCCG Årsrapport 2015, www.dccg.dk). Based on these data and according to the inclusion criteria, 47 patients are eligible candidates per year, and the expected accrual of 60 patients (see below) is two years.

ELIGIBILITY:
Inclusion Criteria:

* Radically resected colon cancer patients with adeno- or signet ring cell carcinomas with high-risk tumors defined as: perforated / pT4NanyM0 (UICC 8th edition) / pTanyNanyM1 with radically resected PM including ovarian metastases
* Performance status 0-1
* Fertile women must use approved contraceptives (see below)
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Radiologically or clinically proven relapse.
* Previous cytoreductive surgery (CRS) with HIPEC
* Other malignant diagnosis within the last 2 years
* Contraindications to laparoscopy (e.g. severe adhesions, peritonitis)
* A history of allergic reaction to oxaliplatin or other platinum containing compounds
* Renal impairment, defined as GFR < 50 ml/min, (Cockcroft-Gault Equation).
* Myocardial insufficiency, defined as NYHA class > 2.
* Impaired liver function defined as bilirubin ≥ 1.5 x UNL (upper normal limit).
* Inadequate haematological function defined as ANC ≤ 1.5 x 109/l and platelets ≤ 100 x 109/l.
* Any other condition or therapy, which in the investigator's opinion may pose a risk to the patient or interfere with the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients with peritoneal recurrence | 3 years
  Based on contrast enhanced CT of the thorax and abdomen 36 months after resection of high-risk colon cancer.

SECONDARY OUTCOMES:
The number of conversions from positive to negative peritoneal lavage cytology | 5 weeks
  Peritoneal lavage cytology will be performed during each PIPAC treatment in order to detect free intraperitoneal tumor cells. Interval of 5 weeks between each PIPAC.
Number of patients where the planned PIPAC procedures are completed | 5 weeks
  Two PIPAC procedures are planned.
Number of patients with treatment related toxicity or complications | 3 months
  Based on CTCAE (vers. 4.0) and Dindo-Clavien´s surgical complications assessment.
1- and 2-year peritoneal recurrence free survival | 2 years
  Based on CT of the thorax and abdomen performed 12- and 24 months after primary resection
1-, 2- and 3-year recurrence free survival, | 3 years
  Based on CT of the thorax and abdomen performed 12-, 24 and 36 months after primary resection
1-, 3- and 5-year overall survival rate | 5 years
  Based on the Danish Civil Registration System

CONTACTS AND LOCATIONS:
Overall Officials: Martin Graversen, MD, Principal Investigator — Odense PIPAC Center
Locations (1):
- Odense PIPAC Center, Department of Surgery, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
The database will be used for publications and presentations by the study group.

REFERENCES:
- [Background] van Gestel YR, de Hingh IH, van Herk-Sukel MP, van Erning FN, Beerepoot LV, Wijsman JH, Slooter GD, Rutten HJ, Creemers GJ, Lemmens VE. Patterns of metachronous metastases after curative treatment of colorectal cancer. Cancer Epidemiol. 2014 Aug;38(4):448-54. doi: 10.1016/j.canep.2014.04.004. Epub 2014 May 17. PMID 24841870
- [Background] Solass W, Kerb R, Murdter T, Giger-Pabst U, Strumberg D, Tempfer C, Zieren J, Schwab M, Reymond MA. Intraperitoneal chemotherapy of peritoneal carcinomatosis using pressurized aerosol as an alternative to liquid solution: first evidence for efficacy. Ann Surg Oncol. 2014 Feb;21(2):553-9. doi: 10.1245/s10434-013-3213-1. Epub 2013 Sep 5. PMID 24006094
- [Background] Demtroder C, Solass W, Zieren J, Strumberg D, Giger-Pabst U, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy with oxaliplatin in colorectal peritoneal metastasis. Colorectal Dis. 2016 Apr;18(4):364-71. doi: 10.1111/codi.13130. PMID 26400556
- [Derived] Graversen M, Detlefsen S, Fristrup C, Pfeiffer P, Mortensen MB. Adjuvant Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) in resected high-risk colon cancer patients - study protocol for the PIPAC-OPC3 Trial. A prospective, controlled phase 2 Study. Pleura Peritoneum. 2018 Jun 12;3(2):20180107. doi: 10.1515/pp-2018-0107. eCollection 2018 Jun 1. PMID 30911655